CLINICAL TRIAL: NCT05391243
Title: Performance of Large Loop Excision of the Transformation Zone (LLETZ) in Women with Cervical Dysplasia in the Follicular Phase Versus the Luteal Phase of the Menstrual Cycle: a Prospective Randomized Trial
Brief Title: Large Loop Excision of the Transformation Zone During Follicular Vs. Luteal Phase of the Menstrual Cycle (LLETZ-MC)
Acronym: LLETZ-MC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Director, Department of Obstetrics and Gynecologiy, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLETZ-MC-1
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cervical Dysplasia
Keywords: cervical dysplasia; LLETZ; LEEP; conization; menstrual cycle
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Conization

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial with 2 groups (follicular phase, luteal phase)
Who Masked: Care Provider
Masking Description: Surgeons will not be provided information about the menstrual cycle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Follicular phase (Other): LLETZ performed during the follicular phase of the menstrual cycle
  Interventions: Procedure: LLETZ
- Luteal phase (Other): LLETZ performed during the luteal phase of the menstrual cycle
  Interventions: Procedure: LLETZ

INTERVENTIONS:
Procedure: LLETZ — Large loop excision of the transformation zone
  Other Names: LEEP; conization

SUMMARY:
Cervical cancer is one of the most common cancers in women and one of the leading causes of death in women worldwide. Pre-cancerous lesions (dysplasias) are detected by the preventive smear test at the gynecologist and can thus contribute to a 100% chance of cure if they are clarified by a colposcopic examination as part of the dysplasia consultation and dysplastic lesions are then surgically removed if necessary (conization).

There are few data in the literature on the influence of the menstrual cycle on the bleeding pattern during and after conization. Hormonal variations during the menstrual cycle affect both the extent of blood flow to reproductive organs and hemostasis. In the follicular phase, there is a decrease in local blood flow in the uterus and pelvic organs and an increase in coagulability. Conversely, in the luteal phase there is an increase in local blood supply and a decrease in coagulability. Therefore, it seems reasonable to perform conization in the follicular phase to possibly reduce the extent and incidence of bleeding and bleeding complications. This assumption is supported by clinical observations. For example, there is evidence from other specialties that selection of the timing of surgery, taking into account the menstrual phase, may influence the risk of bleeding. Another factor of interest in menstruation-based surgical planning is psychological vulnerability, which may also vary with the menstrual cycle. Until now, consideration of the menstrual cycle in surgical planning for conization has not been standard practice and there is no recommendation in this regard in the current S3 guideline of the German Society of Gynecology and Obstetrics.

Therefore, this study now aims to answer the question under prospective randomized conditions whether LLETZ conization performed during the follicular phase results in lower blood loss and higher patient satisfaction and lower anxiety scores compared to LLETZ conization performed during the luteal phase.

DETAILED DESCRIPTION:
HPV and dysplasia of the uterine cervix

Human papillomaviruses (HPV) are the most common sexually transmitted pathogens worldwide. The prevalence in both male and female populations is high. Epidemiological estimates suggest that 85-91% of sexually active adults acquire at least one genital HPV infection by the age of 50, with approximately 95% of HPV infections being spontaneously eliminated within 2 years in terms of HPV immunological clearance. HPV preferentially infects the epithelial cells of the anogenital area and, through incorporation of HPV DNA into the host genome of the basal cells of the squamous epithelium of the cervix and subsequent expression of viral components, causes dysplastic changes in the cervical epithelium that, if left untreated, can develop into invasive carcinoma of the cervix (cervical carcinoma). Cervical carcinoma is the fourth most common cancer as well as the fourth leading cause of cancer-related death in women worldwide, responsible for 6.6% (570,000) of all new cancer cases and 7.5% (311,000) of cancer-related deaths in women in 2018. The precursor of squamous cell carcinoma of the uterine cervix (approximately 80% of all cervical cancers) is cervical intraepithelial neoplasia (CIN), which has three grades of expression (CIN1, CIN 2, and CIN 3). Compared with invasive cervical carcinoma, the incidence of precancerous lesions of the cervix uteri is much higher. It is estimated that approximately 100,000 women in Germany develop high-grade dysplasia (CIN2/CIN3) each year.

Therapy of cervical dysplasia

Dysplasia of the cervix is typically detected during the gynecological screening examination at the gynecologist. Smears are taken from the ectocervix and endocervix and cytologically evaluated for dysplastic cells and smear quality after Papanicolaou staining. For further clarification of dysplastic changes, presentation to a specialized dysplasia consultation is recommended in the case of abnormalities with suspected presence of cervical dysplasia. Histological confirmation of abnormal areas is performed during colposcopic examination. The histopathological processing of the tissue samples and the colposcopic image of the spread of the changes in the cervix then allow individualized therapy planning.

Conization as the standard of surgical treatment

If precancerous lesions with the potential to develop into an invasive cervical tumor are detected, conization (= surgical removal of a cone of tissue from the cervix) is the method of choice for removing the diseased tissue. The worldwide standard surgical procedure for conization is LLETZ conization (="Large Loop Excision of the Transformation Zone"). In addition to the risk of local persistence of precancerous lesions if cervical dysplasia is incompletely removed, LLETZ also increases the risk of preterm delivery in subsequent pregnancy. This risk increases with increasing volume of removed tissue. To reduce or avoid the aforementioned complications, conization should be performed under colposcopic vision and as little healthy cervical tissue as possible should be removed.

Influence of the menstrual cycle on the bleeding pattern during and after conization

Hormonal variations during the menstrual cycle influence both the extent of blood flow to reproductive organs and hemostasis. Concentrations of fibrinogen, von Willebrand factor antigen, and von Willebrand factor activity show significant menstrual cycle variations with maximum values during the luteal phase. In this sense, during the first cycle phase, the follicular phase, there is a decrease in local blood flow in the uterus and pelvic organs and an increase in coagulability. In contrast, in the second cycle phase, the luteal phase, there is a subsequent increase in local blood supply and a decrease in coagulability. Therefore, it seems reasonable to perform conization in the follicular phase to possibly reduce the extent and incidence of bleeding and bleeding complications. This assumption is supported by clinical observations. For example, there is evidence from other specialties that selecting the timing of surgery, taking into account the menstrual phase, may influence the risk of bleeding. In two non-controlled, retrospective studies of patients undergoing mammary reduction surgery and rhinoplasty, the magnitude of intraoperative and postoperative blood loss was lower during the follicular phase than during the luteal phase. In addition, a small randomized trial of 73 patients undergoing cervical uterine surgery (loop electrosurgical excision procedure [LEEP]) found a demonstrable advantage in terms of intraoperative and postoperative blood loss when LEEP was performed during the follicular phase. Another factor of interest in menstruation-oriented surgical planning is psychological vulnerability, which also varies with the menstrual cycle. This factor, which is important for the extent of psychological stress and processing of surgery, also seems to be relevant in the context of conization. Thus, Paraskevaidis et al. were able to show in a randomized study that women who underwent LLETZ conization in the luteal phase had significantly higher anxiety scores and evaluated the surgery more negatively than women who underwent surgery during the follicular phase. This aspect also supports the usefulness of performing conization during the follicular phase. So far, consideration of the menstrual cycle in surgical planning of conization is not standard and there is no recommendation in this regard in the current S3 guideline of the German Society of Gynecology and Obstetrics (DGGG). To date, the selection of the appropriate time for surgery depends only on the patient's time preference and the availability of the surgical site.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Regular menstrual cycle, defined as an interval between 21 and 35 days and a bleeding duration between 3 and 10 days during the last 3 months
* Colposcopy performed preoperatively
* Histologically (by previously performed colposcopy) confirmed dysplasia (CIN 1, CIN 2 or CIN 3)
* Suspicion of low-grade or high-grade squamous intraepithelial lesion based on Papanicolaou smear with inconclusive colposcopy and need for surgical workup to exclude lesions
* Age >18 years

Exclusion Criteria:

* Pregnant patients
* Patients with insufficient knowledge of the German language
* Pre-existing oncological diseases
* Blood coagulation disorders
* Taking blood thinning substances
* Use of a hormonal intrauterine device (e.g. Mirena);
* Use of a progesterone pill or progesterone injectate;
* Use of long cycle contraceptive (no monthly bleeding).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss (weight) | During surgery
  The intraoperative blood loss, measured by the net-weight (in grams) of the surgical swabs used for hemostasis

SECONDARY OUTCOMES:
Intraoperative blood loss (Hb) | Day of surgery
  The intraoperative blood loss, assessed through the difference between the Hb values measured preoperatively and 2 hours postoperatively, respectively.
Intraoperative blood loss (subjective) | Immediately after surgery
  The extent of intraoperative blood loss estimated by the surgeon (blinded to menstrual cycle phase) using a subjective categorization (mild, moderate, severe).
Postoperative bleeding (subjective) | Interview 14 days after surgery
  The extent of postoperative bleeding during the first 24 hours after surgery (assessed by the patient using an 11-item Numerical Rating Scale; 0 [minimal bleeding] - 10 [strong bleeding]).
Postoperative bleeding (days) | Interview 14 days after surgery
  The number of postoperative days where bleeding occurred
Patient's anxiety | On the day of surgery, before surgery
  The patient's anxiety level due to surgery as measured by the Spielberger State-Trait Anxiety Inventory (STAI, situational anxiety STAI-S, trait anxiety, STAI-T). Score range 20 to 80 points for each of the two parts of the test (a higher score means higher levels of anxiety).
Rate of complications | During surgery up to 14 days post surgery
  The occurring intra- and postoperative complications in a period within 14 days after surgery
Cone mass | During surgery, immediately after the excision
  The weight of the cone specimen (measured in grams in the unfixed state)
Procedure duration | At surgery
  Duration of the procedure (from start until complete hemostasis is achieved)
Patient satisfaction | At discharge and 14 days after surgery
  Overall patient satisfaction (11-item numerical rating scale).

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B. Tempfer, MD, MBA, Principal Investigator — Ruhr-Universität Bochum / Marien Hospital Herne
Locations (1):
- Marien Hospital Herne, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request made to the corresponding author. This includes individual participant data underlying the results presented here, after deidentification, as well as data dictionaries and the the study protocol. Data is available after publication, without a specific end date. Requesting investigators must show that their proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication of the study results, no time limit.
Access Criteria: Reasonable request, approval of the intended study by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Workowski KA, Bachmann LH, Chan PA, Johnston CM, Muzny CA, Park I, Reno H, Zenilman JM, Bolan GA. Sexually Transmitted Infections Treatment Guidelines, 2021. MMWR Recomm Rep. 2021 Jul 23;70(4):1-187. doi: 10.15585/mmwr.rr7004a1. PMID 34292926
- [Background] Chesson HW, Dunne EF, Hariri S, Markowitz LE. The estimated lifetime probability of acquiring human papillomavirus in the United States. Sex Transm Dis. 2014 Nov;41(11):660-4. doi: 10.1097/OLQ.0000000000000193. PMID 25299412
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Kuhn W. [Colposcopy in the diagnosis of early cervical cancer]. Pathologe. 2011 Nov;32(6):497-504. doi: 10.1007/s00292-011-1480-9. German. PMID 21984389
- [Background] Mathevet P, Chemali E, Roy M, Dargent D. Long-term outcome of a randomized study comparing three techniques of conization: cold knife, laser, and LEEP. Eur J Obstet Gynecol Reprod Biol. 2003 Feb 10;106(2):214-8. doi: 10.1016/s0301-2115(02)00245-2. PMID 12551795
- [Background] Bevis KS, Biggio JR. Cervical conization and the risk of preterm delivery. Am J Obstet Gynecol. 2011 Jul;205(1):19-27. doi: 10.1016/j.ajog.2011.01.003. Epub 2011 Feb 23. PMID 21345402
- [Background] Jin G, LanLan Z, Li C, Dan Z. Pregnancy outcome following loop electrosurgical excision procedure (LEEP) a systematic review and meta-analysis. Arch Gynecol Obstet. 2014 Jan;289(1):85-99. doi: 10.1007/s00404-013-2955-0. Epub 2013 Jul 11. PMID 23843155
- [Background] Khalid S, Dimitriou E, Conroy R, Paraskevaidis E, Kyrgiou M, Harrity C, Arbyn M, Prendiville W. The thickness and volume of LLETZ specimens can predict the relative risk of pregnancy-related morbidity. BJOG. 2012 May;119(6):685-91. doi: 10.1111/j.1471-0528.2011.03252.x. Epub 2012 Feb 14. PMID 22329499
- [Background] Shaco-Levy R, Eger G, Dreiher J, Benharroch D, Meirovitz M. Positive margin status in uterine cervix cone specimens is associated with persistent/recurrent high-grade dysplasia. Int J Gynecol Pathol. 2014 Jan;33(1):83-8. doi: 10.1097/PGP.0b013e3182763158. PMID 24300540
- [Background] Preaubert L, Gondry J, Mancini J, Chevreau J, Lamblin G, Atallah A, Lavoue V, Caradec C, Baldauf JJ, Bryand A, Henno S, Villeret J, Agostini A, Douvier S, Jarniat A, Riethmuller D, Mendel A, Brun JL, Rakotomahenina H, Carcopino X. Benefits of Direct Colposcopic Vision for Optimal LLETZ Procedure: A Prospective Multicenter Study. J Low Genit Tract Dis. 2016 Jan;20(1):15-21. doi: 10.1097/LGT.0000000000000156. PMID 26704328
- [Background] Knol HM, Kemperman RF, Kluin-Nelemans HC, Mulder AB, Meijer K. Haemostatic variables during normal menstrual cycle. A systematic review. Thromb Haemost. 2012 Jan;107(1):22-9. doi: 10.1160/TH11-07-0481. Epub 2011 Dec 8. PMID 22159564
- [Background] Kadir RA, Economides DL, Sabin CA, Owens D, Lee CA. Variations in coagulation factors in women: effects of age, ethnicity, menstrual cycle and combined oral contraceptive. Thromb Haemost. 1999 Nov;82(5):1456-61. PMID 10595638
- [Background] Andersson O, Blomback M, Bremme K, Wramsby H. Prediction of changes in levels of haemostatic variables during natural menstrual cycle and ovarian hyperstimulation. Thromb Haemost. 1997 May;77(5):901-4. PMID 9184400
- [Background] Sariguney Y, Demirtas Y, Findikcioglu F, Ayhan S, Latifoglu O, Cenetoglu S, Celebi C. Proper timing of breast reduction during the menstrual cycle. Ann Plast Surg. 2004 Dec;53(6):528-31. doi: 10.1097/01.sap.0000134753.15282.cd. PMID 15602247
- [Background] Findikcioglu K, Findikcioglu F, Demirtas Y et al. (2009) Effect of the menstrual cycle on intraoperative bleeding in rhinoplasty patients. Eur J Plast Surg(32): 77e81
- [Background] Gungorduk K, Ozdemir A, Sahin O. Optimal timing of the loop electrosurgical excision procedure according to different phases of the menstrual cycle. J Gynecol Obstet Hum Reprod. 2021 May;50(5):101888. doi: 10.1016/j.jogoh.2020.101888. Epub 2020 Aug 16. PMID 32814158
- [Background] Paraskevaidis E, Davidson EJ, Koliopoulos G, Alamanos Y, Lolis E, Martin-Hirsch P. Bleeding after loop electrosurgical excision procedure performed in either the follicular or luteal phase of the menstrual cycle: a randomized trial. Obstet Gynecol. 2002 Jun;99(6):997-1000. doi: 10.1016/s0029-7844(02)02003-3. PMID 12052589
- See also: German S3 Guidelines — https://www.leitlinienprogramm-onkologie.de/leitlinien/zervixkarzinom-praevention/